CLINICAL TRIAL: NCT02104557
Title: POST MARKETING SURVEILLANCE TO OBSERVE SAFETY AND EFFICACY OF SAYANA(REGISTERED) USED FOR CONTRACEPTION AND MANAGEMENT OF ENDOMETRIOSIS-ASSOCIATED PAIN
Brief Title: Post Marketing Surveillance Study For Sayana®
Acronym: SAYANA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6791036
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Product Surveillance, Postmarketing
Keywords: Sayana; Pregnancy; Contraception; Endometriosis-associated pain; PMS; Post Marketing Surveillance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- prevention of pregnancy: Non intervention
  Interventions: Other: Non intervention
- management of endometriosis-associated pain: Non intervention
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — Non intervention
  Groups: prevention of pregnancy
Other: Non intervention — Non intervention
  Groups: management of endometriosis-associated pain

SUMMARY:
Post Marketing Surveillance To Observe Safety And Efficacy Of Sayana® Used For Contraception And Management Of Endometriosis-Associated Pain

DETAILED DESCRIPTION:
Post Marketing Surveillance required by Korea MFDS regulation. Select among patients who randomly visit the site who meet the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

- Subjects or legally authorized representatives of pediatric subjects agree to provide written informed consent form (ie, data privacy statement).

2.Women subjects who are initiating treatment with Sayana® for the first time as per the local product document for usage

Exclusion Criteria:

* Known or suspected pregnancy.
* Undiagnosed vaginal bleeding.
* Known or suspected malignancy of breast.
* Active thrombophlebitis, or current or past history of thromboembolic disorders, or cerebral vascular disease.
* Significant liver disease.
* Known hypersensitivity to medroxyprogesterone acetate or any of its other ingredients.
* Women who are before menarche or who are post-menopausal.
* Treatment with any investigational agent or device within 30 days prior to the enrollment visit.

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Women subjects who are initiating treatment with Sayana® for the first time as per the local product document for usage
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- South Korea (19):
  - Inje University Haeundae Paik Hospital, Haeundae-gu, Busan
  - Bundang Cha Medical Center, Seongnam-si, Gyeonggi-do
  - CHA Bundang Medical Center-CHA University, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Soon Chun Hyang University Hospital Seoul, Seoul, Korea
  - Ulsan University Hospital, Ulsan, Korea
  - Min Hyunju Women's Clinic, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Inje University Sanggye Paik Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - CHA Gangnam Medical Center, CHA University, Seoul
  - Roen Clinic, Seoul
  - Nana Clinic, Seoul
  - Avenue Clinic, Seoul

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6791036&StudyName=Post%20Marketing%20Surveillance%20To%20Observe%20Safety%20And%20Efficacy%20Of%20Sayana%28registered%29%20Used%20For%20Contraception%20And%20Management%20Of%20Endometriosis-associated%20Pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were planned to be observed for 6 months from enrolment date but few of them were followed beyond 6 months, up to a maximum of 12 months based on investigators' judgement
Pre-assignment Details: Main objective of this study was to conduct safety analysis of Sayana injection in participants during usual care setting so data for both groups (pregnancy prevention group and endometriosis associated pain group) were combined and presented. For efficacy analysis data was collected separately for both groups.
Groups:
- Sayana: Participants were administered with Sayana (medroxyprogesterone acetate) as part of routine practice in Korean health care centers by accredited physicians per the local product document.
Period: Overall Study
Arm/Group | Sayana
Started | 362
Safety Population | 337
Completed | 185
Not Completed | 177
Not completed — Adverse Event | 24
Not completed — Lost to Follow-up | 34
Not completed — Violated the usage and dosage | 14
Not completed — No longer met inclusion/exclusion criteria | 1
Not completed — Administered Sayana prior to the contract | 1
Not completed — Other | 17
Not completed — Change to other contraception methods | 5
Not completed — Discontinuation due to no pain | 1
Not completed — Withdrawal consent | 2
Not completed — Refusal of administration due to unknown reasons | 69
Not completed — Discontinuation of contraception | 9

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of Sayana.
Arm/Group | Sayana
Number analyzed (Participants) | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.92 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. AEs included both serious and all non-serious adverse events.
Time Frame: Baseline up to a maximum of 12 months
Population: Safety analysis set included all participants who received at least 1 dose of Sayana.
Measure: Count of Participants; unit: Participants
Arm/Group | Sayana
Number analyzed (Participants) | 337
Participants
  AEs | 81
  SAEs | 1

2. Primary Outcome: Number of Participants Discontinued From Study Due to AEs
Description: Participants who discontinued permanently from the study due to AEs are reported. An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship.
Time Frame: Baseline up to a maximum of 12 months
Population: Safety analysis set included all participants who received at least 1 dose of Sayana.
Measure: Count of Participants; unit: Participants
Arm/Group | Sayana
Number analyzed (Participants) | 337
Participants | 22

3. Primary Outcome: Number of Participants Used Concomitant Medications for Treating AEs
Description: Number of participants taking any medications other than Sayana (concomitant medication) to treat AEs are reported.
Time Frame: Baseline up to a maximum of 12 months
Population: Safety analysis set included all participants who received at least 1 dose of Sayana.
Measure: Count of Participants; unit: Participants
Arm/Group | Sayana
Number analyzed (Participants) | 337
Participants | 54

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Laboratory tests included hematology, biochemistry, and urinalysis. Clinical significance was identified by investigators' judgements based on laboratory test results.
Time Frame: Baseline up to a maximum of 12 months
Population: Safety analysis set included all participants who received at least 1 dose of Sayana.
Measure: Count of Participants; unit: Participants
Arm/Group | Sayana
Number analyzed (Participants) | 337
Participants | 0

5. Primary Outcome: Percentage of Participants Who Became Pregnant Over Observation Period
Description: The cumulative percent of participants who became pregnant over observation period was calculated as 100*(1- Kaplan-Meier curve at month 12), where the Kaplan-Meier (KM) method for estimating survival function was applied to time-to-pregnancy.
Time Frame: Baseline up to 12 months
Population: Efficacy analysis set included all participants who received at least 1 dose of Sayana and evaluated for efficacy at least once. Here, "Overall number of participants analyzed" = participants who were administered with Sayana for pregnancy prevention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sayana
Number analyzed (Participants) | 182
percentage of participants | 0 [0 to 0]

6. Primary Outcome: Rate of Pregnancies Per 100 Participant-years of Follow-up
Description: Pregnancies per 100 person-years of follow-up defined as major events, incidence rate was calculated as: 100*(total number of participants with effectiveness endpoint)/(total person-years of participants included in the effectiveness analysis set) where total person-years is equal to (last evaluation date of outcome - first date of administration +1)/365.25 for all participants in the effective analysis set.
Time Frame: Baseline up to 12 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: pregnancies per 100 participant-years
Arm/Group | Sayana
Number analyzed (Participants) | 182
pregnancies per 100 participant-years | 0 [0 to 0]

7. Primary Outcome: Change From Baseline in Endometriosis Pain Visual Analogue Scale (VAS) Scores After Administration of First Dose (Month 3) of Study Drug
Description: Participants were asked to indicate the subjective level of endometriosis pain looking back at the last 3 months and mark it with a single vertical mark on the 100 millimeter (mm) horizontal visual analogue scale, where 0 mm represented absence of pain and 100 mm indicated unbearable pain. Higher score indicated more pain. Change from baseline in pain VAS score after administration of first dose of study drug is reported in this outcome measure.
Time Frame: Baseline, Month 3
Population: Efficacy analysis set included all participants who received at least 1 dose of Sayana and evaluated for efficacy at least once. Here, "Overall number of participants analyzed" = participants who were administered with Sayana for the management of endometriosis-associated pain at Month 3.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Sayana
Number analyzed (Participants) | 144
millimeter
  Baseline | 48.32 (31.9)
  Change at Month 3 | -29.63 (29.31)

8. Primary Outcome: Change From Baseline in Endometriosis Pain Visual Analogue Scale (VAS) Scores After Administration of Second Dose (Month 6) of Study Drug
Description: Participants were asked to indicate the subjective level of endometriosis pain looking back at the last 3 months and mark it with a single vertical mark on the 100 mm horizontal visual analogue scale, where 0 mm represented absence of pain and 100 mm indicated unbearable pain. Higher score indicated more pain. Change from baseline in pain VAS score after administration of second dose of study drug is reported in this outcome measure.
Time Frame: Baseline, Month 6
Population: Efficacy analysis set included all participants who received at least 1 dose of Sayana and evaluated for efficacy at least once. Here, "Overall number of participants analyzed" = participants who were administered with Sayana for the management of endometriosis-associated pain at Month 6.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Sayana
Number analyzed (Participants) | 105
millimeter | -33.02 (30.8)

9. Primary Outcome: Change From Baseline in Endometriosis Pain Visual Analogue Scale (VAS) Scores After Administration of Third Dose (Month 9) of Study Drug
Description: Participants were asked to indicate the subjective level of endometriosis pain looking back at the last 3 months and mark it with a single vertical mark on the 100 mm horizontal visual analogue scale, where 0 mm represented absence of pain and 100 mm indicated unbearable pain. Higher score indicated more pain. Change from baseline in pain VAS score after administration of third dose of study drug is reported in this outcome measure.
Time Frame: Baseline, Month 9
Population: Efficacy analysis set included all participants who received at least 1 dose of Sayana and evaluated for efficacy at least once. Here, "Overall number of participants analyzed" =participants who were administered with Sayana for the management of endometriosis-associated pain at Month 9.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Sayana
Number analyzed (Participants) | 10
millimeter | -37.8 (30.7)

10. Primary Outcome: Change From Baseline in in Endometriosis Pain Visual Analogue Scale (VAS) Scores After Administration of Fourth Dose (Month 12) of Study Drug
Description: Participants were asked to indicate the subjective level of endometriosis pain looking back at the last 3 months and mark it with a single vertical mark on the 100 mm horizontal visual analogue scale, where 0 mm represented absence of pain and 100 mm indicated unbearable pain. Higher score indicated more pain. Change from baseline in pain VAS score after administration of fourth dose of study drug is reported in this outcome measure.
Time Frame: Baseline, Month 12
Population: Efficacy analysis set included all participants who received at least 1 dose of Sayana and evaluated for efficacy at least once. Here, "Overall number of participants analyzed" = participants who were administered with Sayana for the management of endometriosis-associated pain at Month 12.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Sayana
Number analyzed (Participants) | 4
millimeter | -49.25 (29.98)

ADVERSE EVENTS:
Time Frame: Baseline up to a maximum of 12 months
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Arm/Group | Sayana
All-Cause Mortality (participants affected / at risk) | 0/337
Serious Adverse Events (participants affected / at risk) | 1/337
Other Adverse Events (participants affected / at risk) | 80/337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sayana (N=337)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sayana (N=337)
Pelvic pain (General disorders) | 1
Headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Weight increase (Metabolism and nutrition disorders) | 3
Skeletal pain (Musculoskeletal and connective tissue disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 13
Breast pain (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 58
Common cold (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Flushing (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02104557/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT02104557/SAP_001.pdf